CLINICAL TRIAL: NCT01118715
Title: Use of Compression Glove to Prevent Complications After Distal Radius Fractures: a Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impractical to enroll the #s needed for statistical significance; project manager relocated
Sponsor: J&M Shuler (Industry)
Responsible Party: Principal Investigator, Michael Shuler, Hand and Upper Extremity Specialist, J&M Shuler
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DRF-001
Record Dates: First submitted 2010-04-30; First posted 2010-05-07 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Post-traumatic Carpal Tunnel Syndrome; Complex Regional Pain Syndrome; Edema
Keywords: distal radius fracture; post-traumatic carpal tunnel syndrome; complex regional pain syndrome; compression glove; edema glove
MeSH Terms: conditions — Complex Regional Pain Syndromes; Edema; Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compression glove (Experimental): Patients in this group have a compression glove incorporated into their splint for 2 weeks post-op, and wear a glove underneath their cast for 3 weeks. The patient then wears the glove at night after cast removal.
  Interventions: Device: Compression glove
- Control (No Intervention): Patients in this group undergo standard recovery procedures. This includes a splint worn for 2 weeks post-op, followed by a short arm cast worn for the next 3 weeks.

INTERVENTIONS:
Device: Compression glove — A compression glove worn during recovery from distal radius fracture
  Arms: Compression glove

SUMMARY:
Distal radius fractures (DRF) are the most common type of fracture in the human body, and a large proportion of DRFs result in complications. Previously proposed preventive strategies have questionable efficacy and may impose additional risks on the patient. Because many complications secondary to distal radius fractures are associated with excessive swelling, a prophylactic means for edema reduction could dramatically reduce morbidity among this population. A compression glove is a non-invasive, non-pharmacological way to reduce edema. Previous studies have confirmed its utility in edema reduction after hand trauma and among patients with chronic inflammatory conditions, but none have sufficiently investigated the application to patients with distal radius fractures, a population in which this intervention could have a large impact. The investigators propose a randomized controlled trial to evaluate use of a compression glove during recovery among patients who have sustained an unstable distal radius fracture. The investigators hypothesize that patients who wear a compression glove after a distal radius fracture:

* Will experience less edema
* Will demonstrate greater functionality
* Will recover more quickly
* Will have lower incidence rates of carpal tunnel syndrome
* Will have lower incidence rates of complex regional pain syndrome

DETAILED DESCRIPTION:
Patients will be recruited from the principle investigator's practice at Athens Orthopedic Clinic. As the only hand and upper-extremity surgeon in the Athens-Clarke county metro area, principle investigator performs the majority of this type of surgery for patients in Athens and surrounding cities. Therefore, the study population should be largely representative of the target population.

Procedures:

1. Patient Identification: Patient presents with distal radius fracture.

   1. An x-ray is taken to decide whether the fracture requires surgical stabilization.
   2. Unstable distal radius fractures will be based on the following criteria:

1. Radial shortening <5 mm at the DRUJ compared with the contralateral side 2. Radial inclination on the posteroanterior radiographs > 15⁰ 3. Sagittal tilt on the lateral projection between 15⁰ dorsal tilt and 20⁰ volar tilt 4. Intra-articular step-off or gap <2 mm of the radiocarpal joint 5. Articular incongruity <2 mm of the sigmoid notch of the distal radius 2. Screening: Patients whose fracture is unstable will be assessed for eligibility using the aforementioned criteria.

3. Consent and de-identification: Patients who are deemed evaluable based on the eligibility criteria will be asked if they are interested in participating in a research study.

1. Those who are interested will meet with a member of the study team, who will explain the study and answer any questions the patient might have.
2. The participant will be given two (2) copies of the informed consent form and HIPAA authorization form. One copy of each document will be signed and returned to the study team, to be kept in a secure location, and the other copy will be given to the participant for his/her records.
3. Each study participant will be assigned a unique study identification number in order to keep his/her identity anonymous. The participant's name and study ID will be recorded on the first page of the case report form, which is detached and kept in a locked filing cabinet immediately following consent. All subsequent data collection will be recorded on the data collection form at follow-up visits with the principle investigator. Data will be entered into a secure, de-identified database by a member of the study team, using the patient's study ID as an identifier. The database will not contain any information that may be used to identify the patient. 4. Surgery: All fractures will be stabilized by volar plate fixation or closed reduction percutaneous pinning using a distal volar radial locking plate or other appropriate implant. 5. Randomization: To avoid any potential bias on the part of the surgeon, patients will be randomized postoperatively to receive either the investigational (glove) or control (no glove) intervention. Therefore, the surgeon will be blinded to intervention status until after patient enrollment and surgical stabilization. 6. Post-surgery: The wound will be dressed steriley, per standard protocol. Initial sterile cast padding will be placed over sterile dressing. For patients in the investigational group, the compression glove will be applied over cast padding, followed by additional padding and then a splint. Patients in the control group will be dressed identically, with the exception of glove application. The splint will be applied for two weeks post-surgery and removal of the splint and application of a short-arm cast will occur at five weeks post-surgery. Additional post-surgical procedures are as follows:

a. 2 weeks- splint is removed; glove is taken off for edema measurements (investigational group); short- arm cast is applied b. 5 weeks- short-arm cast is removed; patient can continue to wear compression glove on an as-needed basis; patient is given post-operative exercise handout c. 3 months- patients meet with study physician for routine follow-up visit d. 6 months- patients meet with study physician for final follow-up visit; once fully healed, patient is given option of having plates removed 7. Therapy: Patients will be given a handout explaining post-operative exercises to be performed at home during recovery.

1. In addition, participants will attend therapy twice weekly, beginning five weeks from surgery. Duration of therapy will be as-needed at the therapist's discretion. Discharge from therapy will be based on the therapist's assessment that the patient has recovered to the extent that they can continue an exercise program at home.
2. Patients who stop coming to therapy prior to discharge will be contacted by the therapists and asked to provide his/her primary reason for not returning. 8. Outcome assessment: outcomes will be assessed at each of four follow-up visits, occurring two weeks, six weeks, three months, and six months from surgery. These coincide with regular post-operative visits, so as to minimize loss to follow-up. Each visit will assess each of the outcome measurements explained in later sections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Between the ages of 18-85
* Patients with unstable unilateral distal radius fractures (requiring surgical stabilization)

Exclusion Criteria:

* Pre-existing cases of carpal tunnel syndrome and/or complex regional pain syndrome
* Nerve or tendon laceration
* Decompression of carpal tunnel concomitant with surgical stabilization
* Additional fractures, including carpal fractures, more proximal fractures of the radius, and finger injuries will be excluded from the study (Ulnar styloid and ulnar head and neck fractures will be included)
* Uncontrolled rheumatoid arthritis patients
* Bilateral fractures
* Unable or unwilling to provide written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-04; Primary Completion 2015-12 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Shuler, MD, Principal Investigator — J&M Shuler
Locations (1):
- Athens Orthopedic Clinic, Athens, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The initial protocol had 94 participants. Analysis was run, however, numbers were trending but not significant. Additional participants were then enrolled to increase the power of the study, leading to a larger participant number(128) than the study originally intended to have.
  There is no intention to continue enrolling subjects.
Period: Overall Study
Arm/Group | Compression Glove | Control
Started | 68 | 60
Completed | 68 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The initial protocol had 94 participants. Analysis was run, however, numbers were trending but not significant. Additional participants were then enrolled to increase the power of the study, leading to a larger participant number(128) than the study originally intended to have.
Groups:
- Total: Total of all reporting groups
Arm/Group | Compression Glove | Control | Total
Number analyzed (Participants) | 68 | 60 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (19.9) | 59.6 (15.3) | 58.22 (18.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 46 | 103
  Male | 11 | 14 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Injured wrist [Count of Participants; unit: Participants]
  Right | 30 | 32 | 62
  Left | 38 | 28 | 66
Pain Scale [Mean (Standard Deviation); unit: units on a scale] — Pain was measured on a Numerical Rating Scale (NRS) which has a minimum score of 0 and a maximum score of 10. The scale appears as a line with 11 equally spaced tick marks on it that are respectively labeled 0-10. Zero indicates 'No Pain,' 5 indicates 'Moderate Pain,' and 10 indicates 'Worst Possible Pain.' The instructions accompanying the scale read, "On a scale of 1-10 what number would you rate the pain that you are experiencing today?"
  units on a scale | 5.1 (2.7) | 6.21 (12.7) | 5.17 (2.95)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-traumatic Carpal Tunnel Syndrome (CTS) or Complex Regional Pain Syndrome (CRPS)
Description: Confirmed cases of Post-traumatic Carpal Tunnel Syndrome (CTS) or Complex Regional Pain Syndrome (CRPS)
Time Frame: 2 wks-24 wks
Population: 'Number Analyzed' is broken down by group (Glove/No Glove) and time frame (2-24 weeks). The overall number of participants analyzed is not consistent with numbers provided in the participant flow module (total participants=128) because not all participants attended all follow-up appointments.
Measure: Count of Participants; unit: Participants
Groups:
- 2 Weeks: Count of patients with a new CTS or CRPS diagnosis at 2 weeks post-surgery.
- 5 Weeks: Count of patients with a new CTS or CRPS diagnosis at 5 weeks post-surgery.
- 12 Weeks: Count of patients with a new CTS or CRPS diagnosis at 12 weeks post-surgery.
- 24 Weeks: Count of patients with a new CTS or CRPS diagnosis at 24 weeks post-surgery.
Arm/Group | 2 Weeks | 5 Weeks | 12 Weeks | 24 Weeks
Number analyzed (Participants) | 123 | 116 | 100 | 86
Participants
  No Glove: number analyzed (Participants) | 58 | 56 | 48 | 47
  No Glove: new dx of CTS or CRPS | 0 | 4 | 4 | 0
  No Glove: no new dx of CTS or CRPS | 58 | 52 | 44 | 47
  Glove: number analyzed (Participants) | 65 | 60 | 52 | 39
  Glove: new dx of CTS or CRPS | 0 | 1 | 2 | 0
  Glove: no new dx of CTS or CRPS | 65 | 59 | 50 | 39

2. Secondary Outcome: Edema
Description: Circumference of Wrist/Finger by Glove or No Glove
Time Frame: 2 wks- 24 weeks
Population: The overall number of participants analyzed is not consistent with numbers provided in the participant flow module (total participants=128) because not all participants attended all follow-up appointments. In addition, QAQC uncovered several cases of appointment records with missing or invalid data.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- 2 Weeks: Wrist or finger circumference measured 2 weeks after surgery.
- 5 Weeks: Wrist or finger circumference measured 5 weeks after surgery.
- 12 Weeks: Wrist or finger circumference measured 12 weeks after surgery.
- 24 Weeks: Wrist or finger circumference measured 24 weeks after surgery.
Arm/Group | 2 Weeks | 5 Weeks | 12 Weeks | 24 Weeks
Number analyzed (Participants) | 99 | 97 | 70 | 56
centimeters
  No Glove - Wrist Circumference: number analyzed (Participants) | 49 | 49 | 35 | 30
  No Glove - Wrist Circumference | 18.09 (1.34) | 17.53 (1.36) | 16.98 (1.37) | 16.74 (1.24)
  Glove - Wrist Circumference: number analyzed (Participants) | 50 | 47 | 35 | 26
  Glove - Wrist Circumference | 17.66 (1.46) | 16.98 (1.50) | 16.75 (1.60) | 17.01 (1.56)
  No Glove 1st Finger: number analyzed (Participants) | 49 | 49 | 35 | 30
  No Glove 1st Finger | 6.94 (.61) | 6.84 (.59) | 6.59 (.56) | 6.50 (.44)
  Glove 1st Finger: number analyzed (Participants) | 50 | 48 | 35 | 26
  Glove 1st Finger | 6.61 (.70) | 6.38 (.66) | 6.57 (.68) | 6.62 (.79)
  No Glove 2nd Finger: number analyzed (Participants) | 49 | 49 | 35 | 30
  No Glove 2nd Finger | 6.77 (.64) | 6.67 (.61) | 6.37 (.56) | 6.28 (.41)
  Glove 2nd Finger: number analyzed (Participants) | 50 | 48 | 35 | 26
  Glove 2nd Finger | 6.47 (.72) | 6.20 (.70) | 6.31 (.73) | 6.43 (.83)
  No Glove 3rd Finger: number analyzed (Participants) | 49 | 49 | 35 | 30
  No Glove 3rd Finger | 6.29 (.58) | 6.31 (.62) | 5.99 (.52) | 5.84 (.41)
  Glove 3rd Finger: number analyzed (Participants) | 50 | 48 | 35 | 26
  Glove 3rd Finger | 6.09 (.69) | 5.86 (.69) | 5.85 (.73) | 5.98 (.76)
  No Glove 4th Finger: number analyzed (Participants) | 49 | 49 | 35 | 30
  No Glove 4th Finger | 5.71 (.51) | 5.82 (.53) | 5.58 (.50) | 5.45 (.41)
  Glove 4th Finger: number analyzed (Participants) | 50 | 48 | 35 | 26
  Glove 4th Finger | 5.56 (.68) | 5.46 (.68) | 5.50 (.68) | 5.56 (.71)

3. Secondary Outcome: Range of Motion
Description: Count of participants (by group) that were capable or full extension or flexion at each encounter.
Time Frame: 2 wks-24 wks
Population: The overall number of participants analyzed is not consistent with numbers provided in the participant flow module (total participants=128) because not all participants attended all follow-up appointments. In addition, QAQC uncovered several cases of appointment records with missing or invalid data. Flexion data missing for 3 subjects and extension data missing for 1 subject at 2 wk visit.
Measure: Count of Participants; unit: Participants
Groups:
- 2 Weeks: Count of participants with full flexion/extension at 2 weeks
- 5 Weeks: Count of participants with full flexion/extension at 5 weeks
- 12 Weeks: Count of participants with full flexion/extension at 12 weeks
- 24 Weeks: Count of participants with full flexion/extension at 24 weeks
Arm/Group | 2 Weeks | 5 Weeks | 12 Weeks | 24 Weeks
Number analyzed (Participants) | 98 | 97 | 70 | 56
Participants
  No Glove - Full Flexion: number analyzed (Participants) | 48 | 49 | 35 | 30
  No Glove - Full Flexion | 24 | 25 | 32 | 28
  Glove - Full Flexion: number analyzed (Participants) | 49 | 48 | 35 | 26
  Glove - Full Flexion | 20 | 31 | 34 | 26
  No Glove - Full Extension: number analyzed (Participants) | 49 | 49 | 35 | 30
  No Glove - Full Extension | 45 | 44 | 33 | 29
  Glove - Full Extension: number analyzed (Participants) | 49 | 48 | 35 | 26
  Glove - Full Extension | 44 | 47 | 35 | 26

4. Secondary Outcome: Grip Strength
Description: Grip strength measured using a hand dynamometer at each visit except @ 2-weeks; grip strength was not measured at 2-weeks because of post-op activity restrictions recommended by the treating physician
Time Frame: 5 wks-24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Groups:
- 5 Weeks: Grip strength measured 5 weeks after surgery
- 12 Weeks: Grip strength measured 12 weeks after surgery
- 24 Weeks: Grip strength measured 24 weeks after surgery
Arm/Group | 5 Weeks | 12 Weeks | 24 Weeks
Number analyzed (Participants) | 116 | 100 | 86
kg
  No Glove: number analyzed (Participants) | 56 | 48 | 47
  No Glove | 6.83 (6.14) | 17.79 (9.17) | 20.73 (11.69)
  Glove: number analyzed (Participants) | 60 | 52 | 39
  Glove | 7.39 (6.04) | 18.10 (10.44) | 23.45 (10.28)

5. Secondary Outcome: DASH Score
Description: Disabilities of the Arm, Shoulder and Hand questionnaire (DASH) is 30-item questionnaire designed to quanitfy functional outcomes of the upper extremity and measure symptoms of pain, physical, emotional, and social domains associated with musculoskeletal disorders of the upper limb. Scores can range from 0-100 with 0 indicating NO disability and 100 indicating extreme disability.
Time Frame: 2 wks- 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 2 Weeks: DASH score measured 2 weeks after surgery
- 5 Weeks: DASH score measured 5 weeks after surgery
- 12 Weeks: DASH score measured 12 weeks after surgery
- 24 Weeks: DASH score measured 24 weeks after surgery
Arm/Group | 2 Weeks | 5 Weeks | 12 Weeks | 24 Weeks
Number analyzed (Participants) | 123 | 116 | 100 | 86
score on a scale
  No Glove: number analyzed (Participants) | 58 | 56 | 48 | 47
  No Glove | 58.12 (22.11) | 39.52 (21.18) | 20.51 (17.24) | 11.50 (14.28)
  Glove: number analyzed (Participants) | 65 | 60 | 52 | 39
  Glove | 62.14 (19.75) | 44.98 (22.30) | 16.42 (16.54) | 10.32 (14.53)

6. Secondary Outcome: Pain on Numerical Rating Scale
Description: Assessment of pain using a numerical rating scale of 0-10, where 0=no pain and 10=worst possible pain
Time Frame: 2 wks- 24 wks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 2 Weeks: Level of pain reported 2 weeks after surgery
- 5 Weeks: Level of pain reported 5 weeks after surgery
- 12 Weeks: Level of pain reported 12 weeks after surgery
- 24 Weeks: Level of pain reported 24 weeks after surgery
Arm/Group | 2 Weeks | 5 Weeks | 12 Weeks | 24 Weeks
Number analyzed (Participants) | 123 | 116 | 100 | 86
units on a scale
  No Glove: number analyzed (Participants) | 58 | 56 | 48 | 47
  No Glove | 2.93 (2.03) | 2.42 (2.11) | 1.32 (1.61) | .81 (1.06)
  Glove: number analyzed (Participants) | 65 | 60 | 52 | 39
  Glove | 3.24 (2.31) | 1.75 (1.57) | 1.03 (1.48) | .73 (1.08)

ADVERSE EVENTS:
Arm/Group | Compression Glove | Control
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/60
Other Adverse Events (participants affected / at risk) | 0/68 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No